CLINICAL TRIAL: NCT02870868
Title: Breathing Interventions for Relaxation: Dosing Through Extended Exhale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Alfredo Gamboa, Assoc. Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160817; 1R61AT009340 (NIH)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Healthy Adults; Stress
Keywords: slow breathing; yoga; mind-body practicers
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slow breathing with exhale greater than inhale (Experimental): Participants randomized to slow breathing with prolonged exhale to inhale ratio received progressive increases in expiration relative to inspiration based on initial assessment until they reached a goal breath length or longest comfortable breath. Prior to performing the breathing practice, subjects in this exhale>inhale condition performed the same yoga movements as the exhale-inhale group.
  Interventions: Behavioral: Slow breathing
- Slow breathing with exhale equal to inhale (Experimental): Participants randomized to slow breathing with equal inspiration and expiration received progressive increases in both inspiration and expiration over 4 weeks until they reach a goal breath length or longest comfortable breath. Goal breaths were assigned based on initial breath assessment. Prior to performing the breathing practice, participants performed a few standardized yoga movements. The purpose of movements was to prepare the subject to sit and focus on breathing. Subjects randomized to exhale=inhale will receive progressive increases in both inspiration and expiration until they reach a goal breath length. Goal breaths will be assigned based on initial breath assessment. Prior to performing the breathing practice, subjects will perform a set of standardized breathing practices. The purpose of these few breathing practices is to prepare the subject to sit and focus on breathing.
  Interventions: Behavioral: Slow breathing

INTERVENTIONS:
Behavioral: Slow breathing — Slow breathing techniques from yoga

SUMMARY:
Breathing exercises are categorized as a mind-body practice. One in ten adults in the U.S. use breathing exercises for health purposes. The aim of this project is to examine if different slow breathing has different physiological and psychological effects.

DETAILED DESCRIPTION:
Breathing exercises are categorized as a mind-body practice. One in ten adults in the U.S. use breathing exercises for health purposes. Slow breathing exercises are commonly used for stress reduction. Higher stress is associated with higher cardiovascular risk. Effective and standardized breathing interventions for stress reduction have not been developed or well-studied. For centuries, mind-body practitioners have proposed that, in addition to breathing slowly, extending the length of exhale relative to inhale increases the dose of relaxation. Few studies have tested this belief. The aim of this proposal is to examine if slow breathing while extending the exhale time relative to the inhale time increases physiological and psychological relaxation. The slow breathing exercises to be studied are based on breathing techniques from yoga. This is a12-week study among healthy adults randomized to daily slow breathing exercises of: (1) exhale greater than inhale versus (2) exhale equal to inhale in length. The first aim of the studies will be to compare 12 weeks of slow breathing with exhale greater than inhale on physiological stress as measured through autonomic tone. The second aim will be to compare changes in psychological stress as measured through validated stress and anxiety questionnaires. The final and third aim will be to measure the correlation between changes in physiological and psychological stress. This project will test if specific breathing techniques produce measurable and meaningful differences in stress in both healthy and disease populations. Because stress reduction is considered the major mechanism of mind-body practices, these studies will advance the field of mind-body science.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60 years
* English speaking

Exclusion Criteria:

* Hypertension
* Heart disease: history of coronary artery disease, myocardial infarction, significant valvular disease, or congestive heart failure
* Diabetes
* Renal disease
* Anxiety disorder
* Depression
* Other psychiatric conditions including schizophrenia or bipolar disorder
* Attention-deficit-disorder or Attention-deficit-hyperactivity disorder
* Musculoskeletal condition limiting capacity to perform simple movements such as chronic lower back pain or neck pain
* Pulmonary disorder (asthma, chronic obstructive lung disease, obstructive sleep apnea)
* Smoker
* Currently taking blood pressure medications, oral diabetic medication or insulin
* Current participation in a mind-body practice/program
* Current cancer other than non- melanoma skin cancer
* Regular swimmer
* Plays wind or brass musical instruments

After two weeks during screening period unable to:

* Breathe 8 or less a minute
* Breathe 3 or less breaths a minute
* Practiced less than 3 times a week

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurjeet Birdee, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Slow Breathing With Exhale Greater Than Inhale: Slow breathing performed with time of exhale longer than inhale
- Slow Breathing With Exhale Equal to Inhale: Slow breathing performed with time of exhale equal to inhale
Period: Overall Study
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Started | 49 | 50
Completed | 47 | 49
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 50 | 99
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (9.2) | 41.0 (8.7) | 41.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 45 | 44 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 4 | 10
  White | 34 | 45 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
High Frequency Heart Rate Variability [Mean (Standard Deviation); unit: milliseconds^second] — Population: Erroneous electrocardiographic measurements for spectral analyses
  milliseconds^second
    number analyzed (Participants) | 41 | 35 | 76
    (all) | 399 (355) | 421 (350) | 409 (350)
PROMIS Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — Measure of psychological stress taken at baseline before any study intervention.
  The scale ranges from 0 (no anxiety) to 100 (maximal anxiety). In the normal adult population, the average of the PROMIS Cooperative Group. (2011). Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety score is 50. A higher score correlates with increased anxiety and a lower score correlates with lower anxiety. Population: Missing data
  units on a scale
    number analyzed (Participants) | 47 | 49 | 96
    (all) | 56.2 (4.8) | 56.5 (5.4) | 56.444 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Change in High Frequency Heart Rate Variability
Description: This is a proxy measure of parasympathetic tone. In normal healthy adults, the average value is around 600 ms^2 (miliseconds*miliseconds). In hypertensive adults, the average value is around 100 ms^2. In patients with autonomic failure (who lacks parasympathetic tone), the average value is around 20 ms^2.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Number analyzed (Participants) | 41 | 35
milliseconds^2 | 399 (355) | 421 (350)

2. Primary Outcome: Magnitude of Change in High Frequency Heart Rate Variability
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Number analyzed (Participants) | 40 | 35
milliseconds^2 | 376 (355) | 485 (463)

3. Primary Outcome: Magnitude of Change in High Frequency Heart Rate Variability
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: milliseconds^2
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Number analyzed (Participants) | 37 | 35
milliseconds^2 | 381 (393) | 487 (476)

4. Primary Outcome: Magnitude of Change in PROMIS Anxiety Scale
Description: Measure of psychological stress taken at baseline before any study intervention.
  The scale ranges from 0 (no anxiety) to 100 (maximal anxiety). In the normal adult population, the average of the PROMIS Cooperative Group. (2011). Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety score is 50. A higher score correlates with increased anxiety and a lower score correlates with lower anxiety.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Number analyzed (Participants) | 47 | 49
units on a scale | 56.2 (4.8) | 56.5 (5.4)

5. Primary Outcome: Magnitude of Change in PROMIS Anxiety Scale
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Number analyzed (Participants) | 47 | 49
units on a scale | 52.4 (5.1) | 53.9 (4.4)

6. Primary Outcome: Magnitude of Change in PROMIS Anxiety Scale
Description: as for outcome 4
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
Number analyzed (Participants) | 45 | 48
units on a scale | 52.0 (4.3) | 51.2 (5.6)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Slow Breathing With Exhale Greater Than Inhale | Slow Breathing With Exhale Equal to Inhale
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Slow Breathing With Exhale Greater Than Inhale (N=49) | Slow Breathing With Exhale Equal to Inhale (N=50)
Lightheadedness (Respiratory, thoracic and mediastinal disorders) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT02870868/Prot_SAP_000.pdf